CLINICAL TRIAL: NCT00097045
Title: Phase 2 Study of Omega Interferon Alone or in Combination With Ribavirin in Subjects With Hepatitis C
Brief Title: Omega Interferon Alone or in Combination With Ribavirin in Subjects With Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Biomed 510-CLP-07
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; HCV; Omega Interferon; Interferon; HCV genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — interferon omega 1; Ribavirin

INTERVENTIONS:
Drug: omega interferon
Drug: Ribavirin

SUMMARY:
This study is designed to compare the safety, tolerability and antiviral effects of omega interferon administered alone to omega interferon administered with ribavirin in the treatment of subjects with chronic Hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
Omega interferon is administered subcutaneously daily for up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 years to 64 years
* Signed and dated written informed consent form
* Infection with HCV genotype 1
* Two HCV RNA levels greater than or equal to 100,000 International Units per mL (IU/mL) at least seven days apart within 6 weeks prior to randomization
* One alanine aminotransferase level greater than the upper limit of normal between three months and twelve months prior to randomization
* At least one alanine aminotransferase level greater than the upper limit of normal between three months and twelve months prior to randomization
* For the duration of treatment with study drug for all subjects and for the duration of treatment with study drug plus an additional six months for subjects who take ribavirin, attenuation of the potential of the subject to become pregnant, or to impregnate a sexual partner, by either:

  1. the use of an approved contraceptive method (e.g., IUD, oral contraceptive, or double-barrier method), or
  2. definitive exclusion by surgery, radiation, menopause or vasectomy
* For women of childbearing potential, negative serum Beta HCG pregnancy test within 14 days prior to randomization

Exclusion Criteria:

* Any additional plausible cause for chronic liver disease, including active infection by other viruses known or suspected to cause hepatitis
* Ascites or other current evidence of portal hypertension
* Child-Pugh classification B or C liver disease
* Clinically apparent jaundice or a total bilirubin exceeding 2 mg/dL (Subjects with Gilbert's Syndrome who meet all other inclusion and exclusion criteria may be admitted to the study with a total bilirubin greater than 2 mg/dL)
* Hemoglobin <12 g/dL
* A platelet count of less than 100,000 per mm3
* A total white blood cell count of less than 3,000 per mm3
* An absolute neutrophil count of less than 1,500 per mm3
* Abnormal thyroid function (Subjects requiring thyroid replacement and who have stable, normal thyroid function may be admitted to the study)
* History of significant renal dysfunction
* History of significant or unstable cardiac disease
* Concurrent alcohol abuse or illicit drug use
* Pregnant or lactating women
* Male partners of women who are pregnant
* Prior usage of an interferon
* Concurrent usage of any antiviral therapy, including another interferon, during the study
* Any concurrent infectious disease requiring antimicrobial treatment
* Positive test for human immunodeficiency virus
* Positive test for illicit drugs
* A history of malignancy (except for previously cured squamous cell or basal cell carcinoma)
* Known hypersensitivity to interferons or ribavirin or related compounds
* A concurrent diagnosis of depression that has not been stable for at least 60 days prior to randomization
* Usage of an investigational drug within the 30 days prior to randomization; or the planned usage of an investigational drug other than omega interferon during the course of the current study
* Prior randomization to this study
* Any condition which, at the discretion of the investigator, would render an individual an inappropriate candidate for this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90
Dates: Start 2004-11; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
HCV RNA levels at clinically relevant timepoints

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Smolensk